CLINICAL TRIAL: NCT00961818
Title: Perceptual, Acoustic and Laryngological Analysis of Vocal Techniques Immediate Effect
Brief Title: Immediate Effect Analysis of Vocal Techniques
Status: Completed | Type: Observational
Sponsor: Tuiuti University of Paraná (Other)
Responsible Party: Masters and Doctorate Program in Communication Disorders of the University Tuiuti of Paraná, University Tuiuti of Paraná
Other Study IDs: UTP; CEP-UTP00026/2008
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Voice Disorders
Keywords: Voice; Voice Quality; Voice Training; Evaluation
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this clinical and experimental study was to verify the immediate effect of vocal techniques: vibration, nasal sound and articulation in women without vocal complaints.

DETAILED DESCRIPTION:
Vocal techniques have been used, but few studies had as their aim to effectively verify its use and effect produced in voice and the larynx. The objective of this clinical and experimental study was to verify the immediate effect of vocal techniques: vibration, nasal sound and articulation. Material and method: 32 female subjects with normal to mild dysphonia participated in the research, with ages from 20 to 45 years. All subjects were submitted to realization of vocal techniques of vibration of the lips, articulation and nasal sounds for twenty minutes. The subjects were submitted to record the voice and laryngostroboscopic exams for perceptual analysis and laryngostroboscopic exams before and after the use of vocal techniques.

ELIGIBILITY:
Inclusion Criteria:

* female subjects
* with normal voices or slightly altered voice
* without vocal complaints

Exclusion Criteria:

* subject with altered voices of moderate and severe grades
* with lesions in the vocal folds; fusiform or double gap on the phonation
* subjects with neurological disorders
* subjects who had been treated earlier speech by voice changes and / or surgery in the larynx

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Were included in the study, female subjects with normal voices evidenced by the slightly altered auditory-perceptual analysis, without vocal complaints, aged between 20 and 45 years.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Subjects were submitted to perceptual analysis and laryngostroboscopic exams before and after the use of vocal techniques. | twenty minutes

CONTACTS AND LOCATIONS:
Overall Officials: Eliane C. Pereira, Master, Principal Investigator — Tuiuti of Parana University
Locations (1):
- Tuiuti of Paraná University, Curitiba, Paraná, Brazil